CLINICAL TRIAL: NCT05128097
Title: Development of a Codified Preventive Approach for the Management of the Main Geriatric Risks
Brief Title: Preventive Approach for the Management of the Main Geriatric Risks
Acronym: Ger-e-Tec
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7792
Record Dates: First submitted 2021-10-06; First posted 2021-11-19 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-10

CONDITIONS: Geriatric Syndromes
Keywords: Geriatric syndromes; psycho-behavioral pathologies; undernutrition,; diabetes
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, EHPAD residents are polypathological (cognitive and psycho-behavioral pathologies, undernutrition, IC, diabetes, COPD, IR, etc.) and multi-medicated. From a medical point of view, this implies the need for regular monitoring and a high level of medical or even multidisciplinary expertise for the healthcare team. The objective of the GER-e-TEC ™ project is to provide these complex patients with telemedicine tools allowing protocolized and personalized, non-intrusive monitoring. The GER-e-TEC ™ project more specifically takes into account the significant issues in nursing homes of aging residents with the main geriatric syndromes (fall, undernutrition, cognitive-behavioral disorders, iatropathogeny, etc.) The objective of the work undertaken is to develop a codified preventive approach for the management of the main geriatric risks, in order to avoid the occurrence of an acute decompensation factor in the elderly.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥65 years old)
* Subject hospitalized between June 17, 2019 to November 13, 2019, in the UF 3723 department, of the Medical Clinic B of the University Hospitals of Strasbourg
* Having not expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Impossibility of providing the subject with enlightened information (difficulties in understanding the subject, etc.)
* Subject under guardianship or guardianship
* Subject under safeguard of justice
* Subject in palliative / end of life situation
* Subject in acute emergency situation

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Major subject (≥65 years old) hospitalized between June 17, 2019 to November 13, 2019, in the UF 3723 department, of the Medical Clinic B of the University Hospitals of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective study of the management of the main geriatric risks in the University HÔptaux de Strasbourg | Files analysed retrospectively from from June 17, 2019 to November 13, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel ANDRES, MD, PhD, Principal Investigator — Médecine interne, Diabète, et Maladies Métaboliques - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Médecine interne, Diabète, et Maladies Métaboliques - Hôpitaux Universitaires de Strasbourg, Strasbourg, France